CLINICAL TRIAL: NCT07210866
Title: AN ARTIFICIAL INTELLIGENCE MODEL FOR INTENSIVE CARE LENGTH OF STAY, NEUROLOGICAL OUTCOME AND COSTS ESTIMATION AFTER CARDIOPULMONARY RESUSCITATION: A COHORT STUDY
Status: Not yet recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Nıgar Kangarlı, Uzman Doctor, Bezmialem Vakif University
Other Study IDs: Nkangarli002
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Cost Analysis; Length of ICU Stay; Neurological Outcome
Keywords: machine learning; cardiopulmonary rescucitation; lenght of stay; cost analysis; neurological outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age >18 years patients after successful cardiopulmonary resuscitation observed in reanimation
  Interventions: Other: no physical or medical interventions

INTERVENTIONS:
Other: no physical or medical interventions — Data from patients after successive rescucitaion will be evaluated by machine learning programs.

SUMMARY:
The study aims to overview patients registered to Bezmialem Vakıf University Hospital Intensive Care Unit after successive cardiac arrest resuscitation from October 2010 to September 2025. The goal is to determine length of stay in reanimation, neurological clinical outcome and costs of these patients at discharge from the department. All these data is intended to be evaluated by artificial intelligence to evaluate a predictive model.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* successive cardiopulmonary resuscitation
* at least 1 hour long admission to ICU after Return Of Spontaneous Circulation (ROSC)

Exclusion Criteria:

* age < 18 years
* >80% missing data in patient records
* patients with no ROSC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above 18 years after successful cardiopulmonary resuscitation with ROSC registered at Bezmialem Vakıf University Hospital Intensive care unit from October 2010 to September 2025 will be included in the resesarch.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Machine Learning Python programme | 3 months
  The created database will be analyzed using a machine learning artificial intelligence algorithm with the Python programming language. After processing missing and incomplete data by artificial intelligence, the database will be divided into two parts: model training and model validation. Meaningful data will be selected through model training, and a prediction model will be built based on these data. To increase the interpretability of the prediction model and help users understand how and why certain predictions are made, the SHapley Additive exPlanations (SHAP) algorithm will be used. In machine learning, the SHAP technique is used to interpret the decision-making processes of complex machine learning models.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT07210866/Prot_SAP_000.pdf